CLINICAL TRIAL: NCT05235295
Title: Fluoroscopic vs Ultrasound Guided Sacroiliac (SI) Joint Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Selin Guven Kose, Principal Investigator, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 126/05
Record Dates: First submitted 2022-02-02; First posted 2022-02-11 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Pain, Chronic
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluoroscopic-guided sacroiliac joint injection (Experimental)
  Interventions: Procedure: Flouroscopy-guided sacroiliac joint injection
- Ultrasound-guided sacroiliac joint injection (Active Comparator)
  Interventions: Procedure: Ultrasound-guided sacroiliac joint injection

INTERVENTIONS:
Procedure: Ultrasound-guided sacroiliac joint injection — Using ultrasound the sacral hiatus in transverse position was identified. Then, sliding laterally and cephalad in transverse position, the posterior superior iliac spine and the posterior sacroiliac joint were identified. The needle was advanced toward the posterior joint space from medial to lateral, using an in-plane technique.
  Arms: Ultrasound-guided sacroiliac joint injection
Procedure: Flouroscopy-guided sacroiliac joint injection — Using anterior posterior and contralateral oblique view the posterior joint line and inferior joint margin were identified and a needle was advanced at the point the posterior inferior joint line was most clearly seen.
  Arms: Fluoroscopic-guided sacroiliac joint injection

SUMMARY:
The investigators aimed to evaluate the effectiveness of intra-articular sacroiliac joint injection under fluoroscopy versus ultrasound guidance

ELIGIBILITY:
Inclusion Criteria:

* Low back and/or gluteal pain without radicular extension for more than 3 months
* Tenderness over the SI joint
* Pain score > 3 by Visual Analogue Scale

Exclusion Criteria:

* Malignancy
* Generalized or local infection
* Coagulopathy
* Allergy to drugs to be injected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Reduction in pain | Change from baseline pain score at 3 months
  Pain assessment will be performed using the Visual Analogue Scale (VAS) score (0 = no pain, 10 = the most severe pain felt).

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | Baseline to 3 months post-procedure
  Mean Change from Baseline in functional disability scores based on Oswestry Disability Index. 0% to 20% indicate minimal disability, 21% to 40% indicate moderate disability, 41%-60% indicates severe disability, 61%-80% means crippled and 81%-100% indicates that the patient is either bed-bound or exaggerating his/her symptoms.
Patient satisfaction Questionnaire | baseline to 3 months post-procedure
  Satisfaction was measured on a 1 to 5 scale,Using score: 5-Excellent, 4-Very Good, 3-Good, 2-Fair, and 1-Poor
Quantitative analgesic questionnaire | at 3 months post-procedure
  A tool designed to record patient-reported pain medication use, create scores to quantify and compare it and track changes in analgesic drug use over time. A higher score indicates higher pain medication use
Procedure time | Intraoperative
  Procedure time was measured using a stopwatch. It was defined as the time from the start of the procedure, the initial image was obtained or first probe placement, until the end of the procedure defined as;transforaminal needle placement was seen clearly.

CONTACTS AND LOCATIONS:
Locations (1):
- Diskapi Yildirim Beyazit Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No